CLINICAL TRIAL: NCT04015375
Title: A Multi-center,Double-blind,Randomized,Three-arm,Placebo-controlled,Parallel-group Study, Comparing Dapsone Gel,7.5% (Torrent Pharma) to Aczone® Gel,7.5% and Both Active Treatments to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: Study Comparing Test to Aczone 7.5% and Both to a Placebo Control in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Collaborators: Catawba Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPSG 1812
Record Dates: First submitted 2019-07-06; First posted 2019-07-11 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone; Gels

STUDY DESIGN:
Intervention Model Description: A multi-center, double-blind, randomized, three-arm, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, Randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dapsone gel, 7.5% (Torrent Pharmaceuticals Ltd.) (Experimental): Topical, once daily for 84 days
  Interventions: Drug: Dapsone gel 7.5% (Torrent Pharmaceuticals Ltd)
- ACZONE® (dapsone) gel, 7.5% (Allergan, INC.) (Active Comparator): Topical, once daily for 84 days
  Interventions: Drug: ACZONE® (dapsone) gel, 7.5% (Allergan, INC.)
- Placebo for Dapsone gel 7.5% (Torrent Pharmaceuticals Ltd) (Placebo Comparator): Topical, once daily for 84 days
  Interventions: Other: Placebo for Dapsone gel 7.5% (Torrent Pharmaceuticals Ltd)

INTERVENTIONS:
Drug: Dapsone gel 7.5% (Torrent Pharmaceuticals Ltd) — Topical gel
  Arms: Dapsone gel, 7.5% (Torrent Pharmaceuticals Ltd.)
Drug: ACZONE® (dapsone) gel, 7.5% (Allergan, INC.) — Topical gel
  Arms: ACZONE® (dapsone) gel, 7.5% (Allergan, INC.)
Other: Placebo for Dapsone gel 7.5% (Torrent Pharmaceuticals Ltd) — Topical gel
  Arms: Placebo for Dapsone gel 7.5% (Torrent Pharmaceuticals Ltd)

SUMMARY:
To evaluate the therapeutic effect of Dapsone and Placebo gel in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
A Multicenter, Double Blind, Randomized, Placebo Controlled, Parallel Group study comparing Dapsone to ACZONE Gel and active treatment to a Placebo control in the treatment of Acne Vulgaris

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
2. Subjects who are 18 years of age or older (up to the age of 40 inclusive) must have provided IRB approved written informed consent. Subjects ages 12 to 17 years of age inclusive must have provided IRB approved written assent; this written assent must be accompanied by an IRB approved written informed consent from the Subject's legally acceptable representative (i.e., parent or guardian). In addition, all Subjects or their legally acceptable representatives (i.e., parent or guardian) must sign a HIPAA authorization.
3. Subjects must have a minimum ≥ 25 non-inflammatory lesions (i.e., open and closed comedones) AND ≥ 20 inflammatory lesions (i.e., papules and pustules) AND ≤ 2 nodulocystic lesions (i.e., nodules and cysts), at baseline on the face. For the purposes of study treatment and evaluation, these lesions should be limited to the facial treatment area. All lesions will be counted, including those present on the nose. Subjects may have acne lesions on other areas of the body which will also be excluded from the count, treatment, and the Investigator's Global Assessment (IGA) evaluation (e.g., on the back, chest and arms).
4. Subjects must have a definite clinical diagnosis of acne vulgaris of severity grade 2, 3, or 4 as per the Investigator's Global Assessment (IGA).
5. Subjects must be willing to refrain from using all other topical acne medications or antibiotics during the 12-week treatment period for acne vulgaris, other than the Investigational Product.
6. Female Subjects of childbearing potential (excluding women who are premenarchal, surgically sterilized or postmenopausal for at least 1 year), in addition to having a negative urine pregnancy test, must be willing to use an acceptable form of birth control during the study from the day of the first dose administration to 30 days after the last administration of study drug . For the purpose of this study the following are considered acceptable methods of birth control: oral or injectable contraceptives, contraceptive patches, Depo-Provera® (stabilized for at least 3 months) NuvaRing® (vaginal contraceptive);Implanon™ (contraceptive implant), double barrier methods (e.g. condom and spermicide),Intrauterine Device (IUD), Essure, or abstinence. If a subject who was abstinent becomes sexually active during the study, a 2nd acceptable method of birth control should be documented. A sterile sexual partner is NOT considered an adequate form of birth control. Hormonal contraceptives should not be initiated or changed during the study.
7. All male Subjects must agree to use accepted methods of birth control with their partners, from the day of the first dose administration to 30 days after the last administration of study drug. Abstinence is an acceptable method of birth control. Female partners should use an acceptable method of birth control as described in the above Item Number 6.
8. Subjects must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits.
9. Subjects must be in good health and free from any clinically significant disease, including but not limited to, conditions that may interfere with the evaluation of acne vulgaris. Such conditions include, but are not limited to the following: autoimmune disease, rosacea; seborrheic dermatitis; perioral dermatitis; corticosteroid-induced acne; carcinoid syndrome; mastocytosis; acneiform eruptions caused by make-up, medication, facial psoriasis and facial eczema.
10. Subjects who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to not change make-up brand/type or frequency of use throughout the study.

Exclusion Criteria:

1. Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
2. Subjects with a history of hypersensitivity or allergy to dapsone and/or any of the study medication ingredients and its excipients.
3. Subjects with the presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneiform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).
4. Subjects with excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris.
5. Subjects who have performed wax depilation of the face within 14 days prior to baseline.
6. Subjects who have used within 6 months prior to baseline or use during the study of oral retinoids (e.g. Accutane®), or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
7. Subjects who have used estrogens or oral contraceptives for less than 3 months prior to baseline; use of such therapy must remain constant throughout the study.
8. Subjects who have used any of the following procedures on the face within 1 month prior to baseline or use during the study:

   1. cryodestruction or chemodestruction,
   2. dermabrasion,
   3. photodynamic therapy,
   4. acne surgery,
   5. intralesional steroids, or
   6. X-ray therapy.
9. Subjects who have used any of the following treatments within 1 month prior to baseline or during the study:

   1. systemic steroids,
   2. spironolactone,
   3. systemic antibiotics,
   4. systemic treatment for acne vulgaris (other than oral retinoids, which require a 6-month washout), or
   5. systemic anti-inflammatory agents
10. Subjects who have used any of the following treatments within 2 weeks prior to baseline or during the study:

    1. topical steroids,
    2. topical retinoids,
    3. topical acne treatments including over-the-counter preparations,
    4. topical anti-inflammatory agents, or
    5. topical antibiotics.
11. Subjects who have received radiation therapy and/or anti-neoplastic agents within 90 days prior to baseline.
12. Subjects who have unstable medical disorders that are clinically significant or have lifethreateningdiseases.
13. Subjects who have on-going malignancies requiring systemic treatment will be excluded from study participation. In addition, Subjects who have any malignancy of the skin of the facial area will also be excluded.
14. Subjects who engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold.
15. Subjects who consume excessive amounts of alcohol (greater than two drinks per day) or of drugs of abuse (including, but not limited to, cannabinoids, cocaine and barbiturates).
16. Subjects who have participated in an investigational drug study (i.e., Subjects have been treated with an investigational drug) within 30 days prior to baseline will be excluded from study participation. Subjects who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion.
17. Subjects who have been previously enrolled in this study.
18. Subjects who have had laser therapy, electrodesiccation and phototherapy (e.g., ClearLight®) to the facial area within 180 days prior to study entry.
19. Subjects who have had cosmetic procedures (e.g., facials) which may affect the efficacy and safety profile of the investigational product within 14 days prior to study entry. Cosmetic procedures and facials are prohibited throughout the study.
20. Subjects who currently have or have recently had bacterial folliculitis on the face.
21. Subjects with a baseline irritation score of 3 = severe (marked, intense).
22. Subjects with known G6PD deficiency, or congenital or idiopathic methemoglobinemia.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1150 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-22 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | 12 weeks
  Mean percent change from baseline to week 12 in the inflammatory (papules and pustules) lesion counts
Change in non-inflammatory counts lesion counts | 12 weeks
  Mean percent change from baseline to week 12 in the non-inflammatory (open and closed comedones) lesion counts

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Thompson, MBA, Study Chair — Catawba Research
Locations (13):
- United States (11):
  - Unison Center for Clinical Trials, Sherman Oaks, California
  - MOORE Clinical Research, Inc., Brandon, Florida
  - FXM Clinical Research Miami, Miami, Florida
  - FXM Clinical Research Miramar, Miramar, Florida
  - MOORE Clinical Research, Inc. (S. Tampa Site), Tampa, Florida
  - MOORE Clinical Research, Inc. (Temple Terrace Site), Temple Terrace, Florida
  - Research Institute of Central Florida, Winter Park, Florida
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - PEAK Research, LLC, Upper Saint Clair, Pennsylvania
  - 3A Research, LLC - WEST, El Paso, Texas
  - 3A Research, LLC - EAST, El Paso, Texas
- Belize (2):
  - Dermatology & Skin Surgery Centre/ FXM Research International, Belize City
  - Dr. Moguel's Clinic/ FXM Research International, Belize City

IPD SHARING:
Plan to Share IPD: No